CLINICAL TRIAL: NCT05071833
Title: Effects of Oral Peppermint Supplementation on Cardiometabolic Parameters
Brief Title: Effects of Peppermint Oil in Cardiometabolic Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Lancashire (Other)
Responsible Party: Principal Investigator, Jonathan Sinclair, Professor, University of Central Lancashire
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Peppermint oil cardiometabolic
Record Dates: First submitted 2021-09-28; First posted 2021-10-08 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Cardiometabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — peppermint oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Identical in taste and colour to the supplement juice, but with no peppermint content.
  Interventions: Other: Placebo
- Peppermint oil (Experimental): 50 uL of peppermint oil, which will be diluted with 100 mL of water - taken twice per day.
  Interventions: Dietary Supplement: Peppermint oil.

INTERVENTIONS:
Dietary Supplement: Peppermint oil. — Peppermint oil.
  Arms: Peppermint oil
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Cardiovascular disease, type 2 diabetes mellitus and associated diseases combined are the leading health burden and cause of mortality worldwide; therefore, the necessity for an intervention is paramount. Dietary interventions to improve cardiometabolic health are highly sought after as they possess less risk than pharmacological drugs. Previous non-randomized interventions have shown that oral peppermint may be beneficial in improving cardiometabolic outcomes. However, to date, no research has explored this using a placebo randomized intervention.

Therefore, the primary purpose of the proposed investigation is to test the ability of oral peppermint oil supplementation to improve cardiometabolic parameters in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Between 18 & 65 years
* Non-smoker
* BMI < 30
* Able to give informed consent

Exclusion Criteria:

* Pregnancy
* Diabetes or any other metabolic/ uncontrolled hypertensive conditions
* Food allergies to peppermint
* Habitual consumption of peppermint
* Not regularly taking medication or antioxidant supplements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-11-05 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | Baseline
  Systolic blood pressure - measured using a digital blood pressure monitor
Systolic blood pressure | 20 days
  Systolic blood pressure - measured using a digital blood pressure monitor

SECONDARY OUTCOMES:
Percent bodyfat | Baseline
  Participants percentage composition of fat - measured using bio-electrical impedance
Percent bodyfat | 20 days
  Participants percentage composition of fat - measured using bio-electrical impedance
Waist to hip ratio | 20 days
  Ratio of waist to hip circumference - measured using anthropocentric tape
Waist to hip ratio | Baseline
  Ratio of waist to hip circumference - measured using anthropocentric tape
Resting metabolic rate | Baseline
  Estimated daily calorie usage (Kcal) at rest - obtained using a metabolic cart through indirect calorimetry.
Resting metabolic rate | 20 days
  Estimated daily calorie usage (Kcal) at rest - obtained using a metabolic cart through indirect calorimetry.
Resting utilization of carbohydrates | 20 days
  Percent contribution of carbohydrate to daily calories - at rest - obtained using a metabolic cart through indirect calorimetry.
Resting utilization of carbohydrates | Baseline
  Percent contribution of carbohydrate to daily calories - at rest - obtained using a metabolic cart through indirect calorimetry.
Resting utilization of fats | Baseline
  Percent contribution of fats to daily calories - at rest - obtained using a metabolic cart through indirect calorimetry.
Resting utilization of fats | 20 days
  Percent contribution of fats to daily calories - at rest - obtained using a metabolic cart through indirect calorimetry.
Blood glucose | Baseline
  Capillary blood glucose - mmol/L
Blood glucose | 20 days
  Capillary blood glucose - mmol/L
Triglyceride glucose index | Baseline
  Calculated as the natural logarithm of (blood triglycerides x blood glucose) /2)
Triglyceride glucose index | 20 days
  Calculated as the natural logarithm of (blood triglycerides x blood glucose) /2)
Blood triglycerides | Baseline
  Capillary blood triglycerides - mmol/L
Blood triglycerides | 20 days
  Capillary blood triglycerides - mmol/L
Blood cholesterol (Total, HDL & LDL) | Baseline
  Capillary blood cholesterol - mmol/L
Blood cholesterol (Total, HDL & LDL) | 20 days
  Capillary blood cholesterol - mmol/L
Blood haemoglobin | Baseline
  Capillary blood haemoglobin - g/L
Blood haemoglobin | 20 days
  Capillary blood haemoglobin - g/L
Coop-Wonka chart | Baseline
  Psychological wellbeing - The Coop-Wonka chart is a six item questionnaire with a 1-5 scoring system for each thus the chart has a maximum score of 30 which indicates the lowest possible psychological Wellbeing.
Beck Depression Inventory | Baseline
  Psychological wellbeing - the Beck Depression Inventory is a 21 questionnaire with questions that range in scoring from 0-3, thus the maximum score is 63 which is the highest depression score possible.
Coop-Wonka chart | 20 days
  Psychological wellbeing - The Coop-Wonka chart is a six item questionnaire with a 1-5 scoring system for each thus the chart has a maximum score of 30 which indicates the lowest possible psychological Wellbeing.
Beck Depression Inventory | 20 days
  Psychological wellbeing - the Beck Depression Inventory is a 21 questionnaire with questions that range in scoring from 0-3, thus the maximum score is 63 which is the highest depression score possible.
State Trait Anxiety Inventory | Baseline
  Psychological wellbeing - the state trait anxiety inventory is a 40 item questionnaire with each question having a 1-4 score system, thus the maximum score is 80 which indicates the highest level of anxiety.
State Trait Anxiety Inventory | 20 days
  Psychological wellbeing - the state trait anxiety inventory is a 40 item questionnaire with each question having a 1-4 score system, thus the maximum score is 80 which indicates the highest level of anxiety.
Insomnia Severity Index | 20 days
  Sleep quality - The Insomnia Severity Index is a brief instrument designed to assess the severity of both nighttime and daytime components of insomnia. The Insomnia Severity Index is a 7-item self-report questionnaire yielding a total score ranging from 0 to 28.
Insomnia Severity Index | Baseline
  Sleep quality - The Insomnia Severity Index is a brief instrument designed to assess the severity of both nighttime and daytime components of insomnia. The Insomnia Severity Index is a 7-item self-report questionnaire yielding a total score ranging from 0 to 28.
Pittsburgh Sleep Quality Index | Baseline
  Sleep quality - The Pittsburgh Sleep Quality index, is a questionnaire that consists of 19 self-rated questions, grouped into 7 components. Each component is scored separately, weighted equally on a 0 - 3 scale and the scores of the 7 components are then added to give a global score, which has a range of 0 - 21 with higher scores indicating worse sleep quality.
Pittsburgh Sleep Quality Index | 20 days
  Sleep quality - The Pittsburgh Sleep Quality index, is a questionnaire that consists of 19 self-rated questions, grouped into 7 components. Each component is scored separately, weighted equally on a 0 - 3 scale and the scores of the 7 components are then added to give a global score, which has a range of 0 - 21 with higher scores indicating worse sleep quality.
Epworth Sleepiness Scale | Baseline
  Sleep quality - The Epworth Sleepiness Scale is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3) with a maximum score of 24.
Epworth Sleepiness Scale | 20 days
  Sleep quality - The Epworth Sleepiness Scale is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3) with a maximum score of 24.
Diastolic blood pressure | Baseline
  Systolic and diastolic blood pressure - measured using a digital blood pressure monitor
Diastolic blood pressure | 20 days
  Systolic and diastolic blood pressure - measured using a digital blood pressure monitor

CONTACTS AND LOCATIONS:
Locations (1):
- Jonathan Sinclair, Preston, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided